CLINICAL TRIAL: NCT05519189
Title: Evaluation of the Value of Perianal Infiltration During Thermodestruction of Haemorrhoidal Disease by Radiofrequency
Acronym: RAFAELOCAL
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Centre Hospitalier Departemental Vendee (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: CHD21_0121
Record Dates: First submitted 2022-08-25; First posted 2022-08-29 (Actual); Last update posted 2026-01-21 (Actual); Status verified 2026-01

CONDITIONS: Hemorrhoids
MeSH Terms: conditions — Hemorrhoids | interventions — Ropivacaine

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Peri-anal infiltration of Ropivacaine (Active Comparator)
  Interventions: Drug: Ropivacaine
- Failure to perform peri-anal ropivacaine infiltration (Experimental)
  Interventions: Other: Failure to perform peri-anal ropivacaine infiltration

INTERVENTIONS:
Drug: Ropivacaine — Peri-anal infiltration of Ropivacaine
  Arms: Peri-anal infiltration of Ropivacaine
Other: Failure to perform peri-anal ropivacaine infiltration — Failure to perform peri-anal ropivacaine infiltration
  Arms: Failure to perform peri-anal ropivacaine infiltration

SUMMARY:
Haemorrhoidal disease is a common and benign condition (1). Anatomically, there is an external and internal component. Only internal haemorrhoidal disease is managed by radiofrequency. Different levels of severity of internal haemorrhoidal disease have been defined by the Goligher classification (1). According to the recommendations for clinical practice established by the French National Society of ColoProctology (SNFCP), grade I and II haemorrhoidal disease should be managed instrumentally after failure of medical treatment. Grade III and IV haemorrhoidal disease is an indication for surgical management in the first instance or after failure of instrumental treatments. The standard technique is the Milligan and Morgan procedure (pedicle haemorrhoidectomy) described in 1937 (2). This technique consists of the removal of the 3 internal haemorrhoidal bundles. It remains the most effective but is responsible for postoperative complications, in particular pain, haemorrhage, anal strictures and anal incontinence (3), (4). Less aggressive techniques have been developed (Longo technique, HAL-RAR technique). The Longo technique is a circular stapling haemorrhoidopexy. The haemorrhoidal packets are brought up into the anal canal with the help of a circular aggravating forceps removing a collar of rectal mucosa. This removal of the mucosa also allows the vascularisation of the haemorrhoidal venous network to be interrupted. The HAL- RAR technique is a non-resection technique consisting of arterial ligation of the haemorrhoidal packets in order to interrupt the vascularisation supplying the haemorrhoidal packets. This technique can be performed with or without Doppler guidance. Recently, Renshaw et al. described a technique for coagulation of haemorrhoidal bundles using a radiofrequency probe (5).

This technique has shown satisfactory results and is an interesting option in the management of haemorrhoidal disease (6) with low postoperative pain (7).

In order to limit patients' postoperative pain and reduce their apprehension during defecation episodes, a perianal block has been shown to reduce postoperative pain in patients with a haemorrhoidectomy technique (8,9). In 2019, a prospective randomised trial (10) confirmed the value of this perianal block without a neurostimulator during a haemorrhoidal pack resection procedure. A perianal infiltration of 40 ml of 0.5% Ropivacaine was performed. These 40ml were divided into 4 injections of 10ml each in the left and right antero-lateral position and in the left and right postero-lateral position in relation to the anal margin.

The hemorrhoidal pack resection technique is known to induce postoperative pain. Haemorrhoidal radiofrequency (RAFAELO® procedure) is a new minimally invasive technique that reduces postoperative pain and is usually performed on an outpatient basis (6). Currently, peri-anal infiltration is routinely performed for all haemorrhoidal surgery whether or not there is a haemorrhoidal resection. No studies have evaluated the relevance of maintaining peri-anal infiltration in non-resected haemorrhoidal surgery and in particular during radiofrequency haemorrhoidal packets. In addition, ropivacaine infiltration is not without risks. Local anaesthesia has potential risks for the patient:

* Adverse reaction or hypersensitivity to local anaesthetics and components
* Infection at the injection site or infiltration
* Haematoma at the injection or infiltration site The aim of our study is to demonstrate the non-inferiority of discontinuing perianal infiltration in patients with thermodestructive haemorrhoidal surgery.

ELIGIBILITY:
Inclusion Criteria:

* Major patient
* Patient scheduled to undergo hemorrhoidal thermodestruction surgery (RAFAELO® procedure)
* Patient able to understand the protocol and having given written informed consent to participate in the study
* Patient affiliated to the social security system or entitled to it

Exclusion Criteria:

* Patient < 18 years old
* Patient with previous hemorrhoidectomy surgery (LONGO technique)
* Patient with previous pexy ligation surgery (HAL-RAR technique)
* Patients with known hypersensitivity to local anaesthetics or components
* Patient with a long term (>1 month) analgesic treatment (level II and III)
* Patient participating in another interventional clinical research protocol involving a drug or clinical investigation of a medical device
* Patient who is pregnant, breastfeeding or able to procreate without contraception
* Patient under guardianship, curatorship or deprived of liberty

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 134 (Actual)
Dates: Start 2023-01-10 (Actual); Primary Completion 2025-12-16 (Actual); Study Completion 2026-01-15 (Actual)

PRIMARY OUTCOMES:
Visual Analogue Scale (VAS) of pain | H6 post-op (6 hours after the start of the operation)
  Minimum value = 0 Maximum value = 10

CONTACTS AND LOCATIONS:
Overall Officials: Emeric ABET, Principal Investigator — Centre Hospitalier Départemental Vendée; Farouk DRISSI, Principal Investigator — Nantes University Hospital; Yann REDON, Principal Investigator — Clinique Mutualiste de l'Estuaire
Locations (3):
- France (3):
  - Centre Hospitalier Départemental Vendée, La Roche-sur-Yon
  - Centre Hospitalier Universitaire de Nantes, Nantes
  - Clinique Mutualiste de l'Estuaire, Saint-Nazaire

IPD SHARING:
Plan to Share IPD: No